CLINICAL TRIAL: NCT06952114
Title: A Single Dose Phase I Study to Evaluate the Safety, Tolerability and Preliminary Effectiveness of Stem Cells Lenses in the Chronic Ocular Graft-versus-Host Disease Subjects
Brief Title: A Study of Stem Cells Lenses in the coGVHD Subjects
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Guangdong ProCapZoom Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLKR-SZ018-0-01
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Chronic Ocular Graft-versus-host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stem Cells Lenses group (Experimental): Each subject will wear Stem Cells Lenses for four consecutive days. After a 4-day treatment period, a 14-day follow-up observation period will be conducted to monitor for potential adverse events.
  Interventions: Drug: Stem Cells Lenses

INTERVENTIONS:
Drug: Stem Cells Lenses — Each subject will wear Stem Cells Lenses for four consecutive days. After a 4-day treatment period, a 14-day follow-up observation period will be conducted to monitor for potential adverse events.

SUMMARY:
This study is a single dose, Phase I study to evaluate the safety, tolerability, and preliminary effectiveness of Stem cells Lenses in the coGVHD Subjects. Three subject's enrollments are Expected. Each subject will wear Stem cells Lenses loaded for four consecutive days. After a 4-day treatment period, a 14-day follow-up observation period will be conducted to monitor for potential adverse events.

This study aims to treat patients with chronic ocular graft-versus-host-disease. Currently, there are no approved drugs for the treatment of coGVHD. Three conventional treatments currently available-systemic administrations, topical treatments, and surgical therapies-have various limitations. allo-HSCT involves the transplantation of hematopoietic stem cells from a healthy donor to a recipient with malignant blood diseases such as leukemia to regenerate the hematopoietic and immune systems. A logical strategy for treating the condition directly would involve the administration of UCMSCs. Using UCMSCs to locally modulate donor T cells and prevent them from attacking the ocular surface tissues of the recipient would be a viable approach to the etiological treatment of coGVHD.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years old, including the boundary value, no gender restriction.
2. Subjects diagnosed with coGVHD caused by hematopoietic stem cell transplantation, with at least 3 months post-transplantation.
3. Meet the clinical diagnostic criteria for coGVHD in the eye: presence of at least one of the following symptoms in either eye: 1) Dryness, burning sensation, foreign body sensation, ocular discomfort, or decreased vision. 2) The total score in either eye ≥ 8 in the absence of systemic chronic graft-versus-host-disease (cGVHD) symptoms, or ≥ 6 in the presence of systemic cGVHD symptoms. (Total score = Schirmer's test score + CFS score + OSDI score + conjunctival congestion).
4. Eye-related symptoms treated conventionally for 1 week prior to screening with no improvement or inadequate response (severity not reduced based on the grading scale of coGVHD).
5. Karnofsky Performance Status (KPS) score > 60.
6. Adequate function of important organs: Absolute neutrophil count ≥ 1.0×10^9/L, platelets count ≥ 75×10^9/L, hemoglobin ≥ 10g/dL, bilirubin ≤ 1.5 times the upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the ULN, and serum creatinine ≤ 1.5 times the ULN.
7. Subjects and their partners have no fertility plans from screening to 6 months after the end of the trial and agree to effective non-pharmacological non-drug contraceptive measures during the trial.
8. Willing to participate in the study, understand and sign the ICF.

Exclusion Criteria:

1. Known allergy to any component of the investigational product.
2. Subjects with any unstable or uncontrolled cardiovascular, pulmonary, gastrointestinal, urogenital, coagulation, immunological, endocrine, metabolic, or other medical conditions that the investigator believes will interfere with the study results or endanger the safety of the subjects.
3. Subjects with other ocular diseases at screening:

   1. Other ocular diseases unrelated to coGVHD, such as blepharospasm.
   2. Acute active fungal, bacterial, or viral keratitis or conjunctivitis, or other acute eye infections.
   3. Corneal ulceration.
   4. Glaucoma, cataracts, or other ocular diseases assessed by the investigator to potentially affect efficacy and safety evaluation.
4. Subjects with a history of Stevens-Johnson Syndrome.
5. Subjects with a history of corneal refractive surgery (e.g., LASIK, PRK) or other corneal surgeries.
6. Subjects who have undergone eye surgery within the previous 3 months.
7. Subjects with a history of corneal contact lens wear who cannot remove them during treatment.
8. Inability to understand and complete the OSDI questionnaire.
9. Participation in other clinical trials within 3 months prior to screening.
10. Subjects with systemic diseases or psychiatric histories that the investigator believes may increase the risk to subjects or affect the evaluation of the study results.
11. Positive test results for human immunodeficiency virus antibodies, Treponema pallidum-specific antibodies (syphilis), or positive hepatitis C antibodies, surface antigen of hepatitis B, history of hepatitis B, or positive hepatitis B core antibody, with recent HBV-DNA levels ≥2000IU/mL in the past 3 months.
12. Subjects with a history of solid tumors.
13. Pregnant or lactating women.
14. Subjects deemed unsuitable for participation in this trial by the investigator.
15. Subjects with active infections will not be recruited.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Adverse events | during the treatment period and within 14 days after treament
  Incidence and severity of AEs from subjects receiving administration to Day 18 post-administration

SECONDARY OUTCOMES:
Corneal fluorescein staining scores | From baseline to Day 4 and Day 18 post-administration
  Changes in corneal fluorescein staining scores
Ocular surface disease | From baseline to Day 4 and Day 18 post-administration
  Changes in ocular surface disease index scores
Schirmer's test | From baseline to Day 4 and Day 18 post-administration
  Changes in Schirmer's test
Tear osmolarity | From baseline to Day 4 and Day 18 post-administration
  Changes in tear osmolarity

IPD SHARING:
Plan to Share IPD: No